CLINICAL TRIAL: NCT03581916
Title: An Open-Label Study to Investigate the Total Body Distribution and Radiation Dosimetry of the Positron Emission Tomography Ligand 18F-JNJ-64326067 in Healthy Subjects
Brief Title: A Study to Investigate the Whole Body Distribution and Radiation Dosimetry of the Positron Emission Tomography Ligand Fluoride-18 (18F)-JNJ-64326067 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR108426; 64326067EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-64326067

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-JNJ-64326067 (Experimental): Participants will receive single intravenous (IV) bolus injection of 18F-JNJ-64326067 on Day 1.
  Interventions: Drug: 18F-JNJ-64326067

INTERVENTIONS:
Drug: 18F-JNJ-64326067 — 18F-JNJ-64326067 will be administered intravenously between a dose of 185 Megabecquerel (MBq) to 370 MBq.

SUMMARY:
The purpose of this study is to measure the whole-body distribution and radiation dosimetry of 18F-JNJ-64326067 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy for their age group on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening or Day 1 predose. If there are abnormalities, they must be consistent with the age of the study population. This determination must be recorded in the participant's source documents and initialed by the investigator
* Otherwise healthy for their age group on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Women must be postmenopausal (must be documented by medical records or physician's note). A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level at screening (greater than [>] 40 International Units Per Liter/ milli International Units Per milliLiter [IU/L) or mIU/mL]) in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy, however in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, a man:

  (a) who is sexually active with a woman of childbearing potential and has not had vasectomy must agree to use a barrier method of contraception (that is, condom). In addition, their female partner should also use a highly effective method of birth control (example, hormonal contraception) for at least the same duration, (b) who is sexually active with a woman who is pregnant must use a condom, (c) must agree not to donate sperm
* Willing and able to adhere to the prohibitions and restrictions specified for this clinical study

Exclusion Criteria:

* Radiation exposure through prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 milli sievert (mSv), which would be above the acceptable annual limits established by the United State (US) Federal Guidelines
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, epilepsy or fits or unexplained black outs, or any other illness that the Investigator considers should exclude the participant
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCV) or human immunodeficiency virus (HIV) antibodies at screening
* History of drug or alcohol use disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria within 6 months before screening or positive test result(s) for alcohol and/or drugs of abuse (opiates (including methadone), cocaine, amphetamines, cannabinoids, barbiturates, 3,4-methylenedioxy-methamphetamine (MDMA) and benzodiazepines) at screening or admission
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with written concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Effective Radiation Dose Following Injection of 18F-JNJ-64326067 per Organ | Day 1
  The Effective Dose (ED) per organ will be calculated using Organ Level Internal Dose Assessment (OLINDA) software. After injection of 370 megaBecquerel (MBq) of 18F-JNJ-64326067, a series of whole-body positron emission tomography (PET) images will be obtained over a period of up to 6 hours and corrected for attenuation by computed tomography (CT) transmission scans using PET/CT. The unit of radioactivity will be milli Sieverts per mega Becquerel (mSv/MBq) for each organ and the effective dose per participant. The final values will be averaged across the participants.
Effective Radiation Dose Following Injection of 18F-JNJ-64326067 for Whole Body | Day 1
  The ED for whole body will be calculated using OLINDA software. After injection of 370 MBq of 18F-JNJ-64326067, a series of whole-body PET images will be obtained over a period of up to 6 hours and corrected for attenuation by CT transmission scans using PET/CT. The unit of radioactivity will be mSv/MBq for the whole body and the effective dose per participant. The final values will be averaged across the participants.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 36 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Invicro, New Haven, Connecticut, United States